CLINICAL TRIAL: NCT05838794
Title: Effectiveness of McKenzie Exercises With and Without Stabilization Exercises in Patients With Nonspecific Chronic Neck Pain: A Randomized Controlled Trial
Brief Title: McKenzie Exercises for Chronic Neck Pain: Stabilization vs. Non-Stabilization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ahram Canadian University (Other)
Responsible Party: Principal Investigator, Mohamed Magdy ElMeligie, Lecturer of Physical Therapy and Director of Electromyography Lab, Ahram Canadian University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 012/004222
Record Dates: First submitted 2023-04-19; First posted 2023-05-03 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: Neck Pain; Cervical Pain
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The assessors who will measure the outcomes will be blinded to the group allocation of participants. However, participants and the treating physiotherapist will not be blinded to the group allocation due to the nature of the intervention. Participants will be instructed not to reveal their group allocation to the assessor during the outcome assessment. To ensure blinding, the assessors will be instructed not to ask any questions that may reveal the group allocation of the participants. In addition, the assessors will be instructed not to discuss the study with the participants to avoid any potential unblinding.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mckenzie exercise for neck (Active Comparator): Participants in the McKenzie exercise for neck group will receive a six-week exercise program that includes the McKenzie exercise protocol for neck pain. The program will consist of three 30-45 minute sessions per week, for a total of 18 sessions over six weeks. The exercises will be performed under the supervision of a physiotherapist in the outpatient clinic. The McKenzie exercise protocol for neck pain involves a series of movements that aim to reduce pain and improve range of motion in the cervical spine. The exercises are tailored to each participant's individual needs and may include sustained postures, repeated movements, and mobilization techniques. Participants will be instructed to perform the exercises at home as well, as part of a home exercise program, to ensure that they are performing the exercises correctly and consistently. Participants in this group will not receive any additional stabilization exercises.
  Interventions: Other: Mckenzie exercise for neck
- Mckenzie ex for neck + Stabilization exercise for (Experimental): Participants in the McKenzie exercises for neck with cervical and scapulothoracic stabilization exercises group will receive a six-week exercise program that includes the McKenzie exercise protocol for neck pain and cervical and scapulothoracic stabilization exercises, performed under the supervision of a physiotherapist in the outpatient clinic. The program consists of three 30-45 minute sessions per week for a total of 18 sessions over six weeks. Participants will perform the McKenzie exercise protocol for neck pain first, followed by cervical and scapulothoracic stabilization exercises. Stabilization exercises aim to improve strength, endurance, and neuromuscular control of the cervical and scapulothoracic muscles. Participants will be instructed to perform the exercises at home as part of a home exercise program to ensure proper technique and consistency. This group receives both the McKenzie exercise protocol for neck pain and cervical and scapulothoracic stabilization exercises.
  Interventions: Other: Mckenzie exercise for neck; Other: Stabilization exercise

INTERVENTIONS:
Other: Mckenzie exercise for neck — The McKenzie protocol will be used to manage extension, rotation, and lateral flexion dysfunctions in patients with non-specific neck pain. An experienced physical therapist will perform the protocol 3 times a week for 6 weeks, tailoring exercises to each patient's individual needs based on limited and painful directions of movement. Exercises include retraction, extension, rotation, lateral flexion, and overpressure techniques. Patients will receive education on posture and body mechanics, and exercises will be progressed over time as the patient improves.
Other: Stabilization exercise — Cervical and scapulothoracic stabilization exercises will be performed by an experienced physical therapist 3 times a week for 6 weeks, with each session including a warm-up, stabilization exercises, and cool-down and stretching exercises. Postural education will be provided using mirrors to find a neutral balanced position, and the cervical bracing technique with deep neck flexor activation will be used to stabilize the cervical spine. Upper extremity range of motion exercises and cervical dynamic isometric exercises with elastic resistive bands will also be performed. Scapulothoracic stabilization exercises will include specific exercises for muscles affecting scapular orientation related to neck pain, using latex bands with mild or medium tension.
  Arms: Mckenzie ex for neck + Stabilization exercise for

SUMMARY:
PURPOSE: To compare the effects of mckenzie exercises plus stabilization exercise to those of mckenzie exercises alone on disability, pain, range of motion (ROM) in patients with nonspecific chronic neck pain (NSCNP).

BACKGROUND: Little is known about the efficacy of providing mckenzie exercises in addition to cervical and scapulothoracic stabilization exercises in people with NSCNP.

HYPOTHESES We hypothesize that there will be no significant effect of adding stabilization exercises to mckenzie exercises than mckenzie exercises alone in patients with NSCNP.

RESEARCH QUESTION: Is there a statistically significant effect of adding stabilization exercises to mckenzie exercises on outcomes of patients with NSCNP?

ELIGIBILITY:
Inclusion Criteria:

1. Ages between 30 and 50 years
2. Localized chronic neck pain without an exact etiology
3. Absence of any arm pain or discomfort that could be replicated by neck mobility or irritant assessment
4. Pain exists in the dorsal area, between two horizontal lines: the first line passes through 5) the lower half of the occipital area, and the second line runs through the spinous process of the first dorsal vertebra

Exclusion Criteria:

1. Neck pain caused by any other complications, such as a neoplasm, neurological diseases, or vascular diseases
2. History of neck surgery or fracture
3. Serious medical conditions that could affect participation in the study, such as cardiovascular disease, cancer, or autoimmune disorders
4. Use of medication that could affect neck pain or exercise tolerance, such as opioids, muscle relaxants, or corticosteroids
5. Participation in other treatments or interventions for neck pain during the study period
6. Inability to understand or comply with study procedures or interventions, such as language barriers or cognitive impairment

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 76 (Actual)
Dates: Start 2023-04-21 (Actual); Primary Completion 2023-08-06 (Actual); Study Completion 2023-08-06 (Actual)

PRIMARY OUTCOMES:
Pain intensity via Numeric pain rating scale | Changes in pain intensity at baseline and 6 weeks after end of treatment program.
  The primary outcome measure will be pain intensity, assessed using the Numeric Pain Rating Scale (NPRS). The intervention will consist of a 4-week program of cervical and scapulothoracic stabilization exercises, performed 3 times a week under the supervision of an experienced physical therapist. Pain intensity will be measured at baseline and 6 weeks after the end of the treatment program.

SECONDARY OUTCOMES:
Neck disability index | Changes in disability at baseline and 6 weeks after end of treatment program.
  The Neck Disability Index (NDI) is a standardized questionnaire that assesses the degree of disability related to neck pain. It consists of 10 questions that evaluate the impact of neck pain on daily activities, such as personal care, lifting, reading, driving, and sleeping. Each question is rated on a scale from 0 to 5, with a total score ranging from 0 to 50. Higher scores indicate greater disability related to neck pain. The NDI is a widely used and validated tool for measuring neck pain-related disability and has been shown to be responsive to changes in disability over time. It is a recommended outcome measure in clinical trials and practice guidelines for patients with neck pain.
Cervical range of motion | Changes in cervical range of motion at baseline and 6 weeks after end of treatment program.
  Cervical range of motion will be assessed with the patient sitting comfortably on a chair, with both feet flat on the floor, hips and knees at 90° of flexion, and buttocks positioned against the back of the chair. A cervical range-of-motion (CROM) device will be placed on the top of the head, and the patient will be asked to move the head as far as possible without pain in a standard fashion: flexion, extension, right lateral flexion, left lateral flexion, right rotation, and left rotation. Three trials will be conducted for each direction of movement, and the mean values of the 3 trials will be recorded for analysis. The reliability of the CROM device in previous studies indicates intraclass correlation coefficients ranging from 0.66 to 0.94, suggesting that it is a valid and reliable method for measuring cervical range of motion.

CONTACTS AND LOCATIONS:
Overall Officials: Amal Fawzy, Ph.d, Study Chair — Faculty of Physical Therapy, Ahram Canadian University
Locations (1):
- Outpatient clinic of faculty of physical therapy, Ahram Canadian University, Al Ḩayy Ath Thāmin, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The individual participant data (IPD) collected during this study will be available upon reasonable request. Requests for access to the data should be submitted via email to mohamed.elmeligie@acu.edu.eg. All requests will be reviewed by the study investigators to ensure that they are reasonable and consistent with the ethical principles of the study. Access to the data will be granted in compliance with applicable laws and regulations, and with appropriate safeguards to protect the privacy and confidentiality of study participants.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: During the study and after 1 year of ending the trial
Access Criteria: via email to mohamed.elmeligie@acu.edu.eg